CLINICAL TRIAL: NCT01381328
Title: GePheRal: Clinical Validation of the Genotypic Diagnosis of Hiv-1 Resistance to Raltegravir by Parallel Analysis of the Genotype and Phenotype Profiles of Resistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: IRCCS San Raffaele (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Elisabetta Carini, Professor Massimo Clementi, Università Vita-Salute San Raffaele
Other Study IDs: Gepheral; Merck Sharp & Dohme Corp. (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: HIV-1 Infected Patients; Fold-change Resistance; Resistance Mutations
Keywords: HIV-1 infected patients; RALTEGRAVIR regimen; genotypic evaluations; phenotypic evaluations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RAL Group: HIV-1 infected patients failing to a RALTEGRAVIR-containing regimen

SUMMARY:
The purpose of this study is to correlate the different patterns of resistance mutations observed in vivo in patients failing RAL treatment with the fold-change resistance determined by the phenotypic assay.

DETAILED DESCRIPTION:
The secondary objectives are, as follows:

* to establish standardised genotypic assay for the HIV-1 pol gene region (region of interest, sensitivity, mutations involved as primary or compensatory changes, role of polymorphism present at baseline).
* to reach consensus on the algorithm interpretation of in house ex-vivo genotypic evaluations.
* to assess the genetic changes in RAL-failing patients under continuous drug pressure or drug discontinuation (dynamics of the reversion of resistance mutations).
* to evaluate in RAL resistant HIV-1 variants the changes in replication capacity (RC) (baseline vs. following-timepoints).
* to evaluate the immunological and virological trend associated with a raltegravir-regimen failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years of age) treatment-experienced, HIV-infected subjects of either sex and of any race, failing to a RAL-containing regimen will be enrolled in the study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
- mean value of fold-change resistance determined by the phenotypic assay at baseline | baseline

SECONDARY OUTCOMES:
changes of fold-change resistance determined by the phenotypic assay with respect to baseline. | 24 and 48 hours, W1, W2, W3 and W4 upon discontinuation
genetic changes under continuous drug pressure or drug discontinuation with respect to baseline(dynamics of the reversion of resistance mutations) | 24 and 48 hours, W1, W2, W3 and W4 upon discontinuation.
changes of the replication capacity with respect to baseline | 24 and 48 hours, W1, W2, W3 and W4 upon discontinuation.
changes of HIV-RNA with respect to baseline | 24 and 48 hours, W1, W2, W3 and W4 upon discontinuation
changes in CD4, CD4%, CD8, CD8% with respect to baseline | 24 and 48 hours, W1, W2, W3 and W4 upon discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Clementi, Prof., Principal Investigator — University Vita-Salute San Raffaele Laboratory of Microbiology and Virology; Antonella Castagna, MD, Study Director — Department of Infectious Diseases, IRCCS San Raffaele Hospital
Locations (1):
- Department of Infectious Diseases, IRCCS San Raffaele Hospital, Milan, Italy

REFERENCES:
- [Background] Engelman A, Mizuuchi K, Craigie R. HIV-1 DNA integration: mechanism of viral DNA cleavage and DNA strand transfer. Cell. 1991 Dec 20;67(6):1211-21. doi: 10.1016/0092-8674(91)90297-c. PMID 1760846
- [Background] Pommier Y, Johnson AA, Marchand C. Integrase inhibitors to treat HIV/AIDS. Nat Rev Drug Discov. 2005 Mar;4(3):236-48. doi: 10.1038/nrd1660. PMID 15729361
- [Background] Anker M, Corales RB. Raltegravir (MK-0518): a novel integrase inhibitor for the treatment of HIV infection. Expert Opin Investig Drugs. 2008 Jan;17(1):97-103. doi: 10.1517/13543784.17.1.97. PMID 18095922
- [Background] Grinsztejn B, Nguyen BY, Katlama C, Gatell JM, Lazzarin A, Vittecoq D, Gonzalez CJ, Chen J, Harvey CM, Isaacs RD; Protocol 005 Team. Safety and efficacy of the HIV-1 integrase inhibitor raltegravir (MK-0518) in treatment-experienced patients with multidrug-resistant virus: a phase II randomised controlled trial. Lancet. 2007 Apr 14;369(9569):1261-1269. doi: 10.1016/S0140-6736(07)60597-2. PMID 17434401
- [Background] Cooper DA, Steigbigel RT, Gatell JM, Rockstroh JK, Katlama C, Yeni P, Lazzarin A, Clotet B, Kumar PN, Eron JE, Schechter M, Markowitz M, Loutfy MR, Lennox JL, Zhao J, Chen J, Ryan DM, Rhodes RR, Killar JA, Gilde LR, Strohmaier KM, Meibohm AR, Miller MD, Hazuda DJ, Nessly ML, DiNubile MJ, Isaacs RD, Teppler H, Nguyen BY; BENCHMRK Study Teams. Subgroup and resistance analyses of raltegravir for resistant HIV-1 infection. N Engl J Med. 2008 Jul 24;359(4):355-65. doi: 10.1056/NEJMoa0708978. PMID 18650513
- [Background] Canducci F, Sampaolo M, Marinozzi MC, Boeri E, Spagnuolo V, Galli A, Castagna A, Lazzarin A, Clementi M, Gianotti N. Dynamic patterns of human immunodeficiency virus type 1 integrase gene evolution in patients failing raltegravir-based salvage therapies. AIDS. 2009 Feb 20;23(4):455-60. doi: 10.1097/QAD.0b013e328323da60. PMID 19165083
- [Background] Nakahara K, Wakasa-Morimoto C, Kobayashi M, Miki S, Noshi T, Seki T, Kanamori-Koyama M, Kawauchi S, Suyama A, Fujishita T, Yoshinaga T, Garvey EP, Johns BA, Foster SA, Underwood MR, Sato A, Fujiwara T. Secondary mutations in viruses resistant to HIV-1 integrase inhibitors that restore viral infectivity and replication kinetics. Antiviral Res. 2009 Feb;81(2):141-6. doi: 10.1016/j.antiviral.2008.10.007. Epub 2008 Nov 21. PMID 19027039
- [Background] Kobayashi M, Nakahara K, Seki T, Miki S, Kawauchi S, Suyama A, Wakasa-Morimoto C, Kodama M, Endoh T, Oosugi E, Matsushita Y, Murai H, Fujishita T, Yoshinaga T, Garvey E, Foster S, Underwood M, Johns B, Sato A, Fujiwara T. Selection of diverse and clinically relevant integrase inhibitor-resistant human immunodeficiency virus type 1 mutants. Antiviral Res. 2008 Nov;80(2):213-22. doi: 10.1016/j.antiviral.2008.06.012. Epub 2008 Jul 14. PMID 18625269
- [Background] Ceccherini-Silberstein F, Malet I, D'Arrigo R, Antinori A, Marcelin AG, Perno CF. Characterization and structural analysis of HIV-1 integrase conservation. AIDS Rev. 2009 Jan-Mar;11(1):17-29. PMID 19290031
- [Background] Malet I, Delelis O, Valantin MA, Montes B, Soulie C, Wirden M, Tchertanov L, Peytavin G, Reynes J, Mouscadet JF, Katlama C, Calvez V, Marcelin AG. Mutations associated with failure of raltegravir treatment affect integrase sensitivity to the inhibitor in vitro. Antimicrob Agents Chemother. 2008 Apr;52(4):1351-8. doi: 10.1128/AAC.01228-07. Epub 2008 Jan 28. PMID 18227187
- [Background] Menzo S, Monachetti A, Balotta C, Corvasce S, Rusconi S, Paolucci S, Baldanti F, Bagnarelli P, Clementi M. Processivity and drug-dependence of HIV-1 protease: determinants of viral fitness in variants resistant to protease inhibitors. AIDS. 2003 Mar 28;17(5):663-71. doi: 10.1097/01.aids.0000050852.71999.5f. PMID 12646788
- [Background] Sichtig N, Sierra S, Kaiser R, Daumer M, Reuter S, Schulter E, Altmann A, Fatkenheuer G, Dittmer U, Pfister H, Esser S. Evolution of raltegravir resistance during therapy. J Antimicrob Chemother. 2009 Jul;64(1):25-32. doi: 10.1093/jac/dkp153. Epub 2009 May 14. PMID 19447792
- [Background] Malet I, Delelis O, Soulie C, Wirden M, Tchertanov L, Mottaz P, Peytavin G, Katlama C, Mouscadet JF, Calvez V, Marcelin AG. Quasispecies variant dynamics during emergence of resistance to raltegravir in HIV-1-infected patients. J Antimicrob Chemother. 2009 Apr;63(4):795-804. doi: 10.1093/jac/dkp014. Epub 2009 Feb 16. PMID 19221102